CLINICAL TRIAL: NCT01680471
Title: Comparative Study on the Effects of Capacities of Midazolam on Delirium After Sevoflurane Anesthesia in Pediatric Strabismus Surgery : a Randomized Double- Blinded Trial
Brief Title: A Study on the Effects of Midazolam on Delirium After Sevoflurane Anesthesia in Pediatric Strabismus Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Korea University Anam Hospital (Other)
Responsible Party: Principal Investigator, Eun Jung Cho, Anesthesiology and Pain Medicine Department, Korea University Anam Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: ECho2012
Record Dates: First submitted 2012-08-28; First posted 2012-09-07 (Estimated); Last update posted 2013-01-04 (Estimated); Status verified 2013-01

CONDITIONS: Child; Anesthesia Morbidity; Delirium on Emergence
Keywords: emergence agitation; midazolam; sevoflurane; strabismus
MeSH Terms: conditions — Emergence Delirium; Strabismus | interventions — Midazolam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Midazolam 0.03mg/kg (Experimental): This group will be injected intravenous midazolam 0.03mg/kg five minutes before the end of surgery.
  Interventions: Drug: Midazolam 0.03mg/kg
- Midazolam 0.05mg/kg (Experimental): This group will be injected intravenous midazolam 0.05mg/kg five minutes before the end of surgery.
  Interventions: Drug: Midazolam 0.05mg/kg
- Placebo (Placebo Comparator): This group will be injected intravenous normal saline five minutes before the end of surgery.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Midazolam 0.03mg/kg — This group will be injected intravenous midazolam 0.03mg/kg five minutes before the end of surgery.
  If emergence agitation is severe, the patients will be treated by psychological support from the parents or nurse and intravenous fentanyl 1㎍/kg.
  Other Names: MIDAZOLAM BUKWANG INJ 5mg/5ml
  Arms: Midazolam 0.03mg/kg
Drug: Midazolam 0.05mg/kg — This group will be injected intravenous midazolam 0.05mg/kg five minutes before the end of surgery.
  If emergence agitation is severe, the patients will be treated by psychological support from the parents or nurse and intravenous fentanyl 1㎍/kg.
  Other Names: MIDAZOLAM BUKWANG INJ 5mg/5ml
  Arms: Midazolam 0.05mg/kg
Drug: Placebo — This group will be injected intravenous normal saline five minutes before the end of surgery.
  If emergence agitation is severe, the patients will be treated by psychological support from the parents or nurse and intravenous fentanyl 1㎍/kg.
  Other Names: NORMAL SALINE INJ(Sodium chloride 9g/1000mL)
  Arms: Placebo

SUMMARY:
Sevoflurane with its rapid induction and emergence, hemodynamic stability, and nonirritating airway properties, has acquired widespread acceptance in children. However, sevoflurane has been reported to be associated with emergence agitation in children, with a reported incidence of up to 80%.

The purpose of this study is to verify that the prophylactic use of midazolam, which is a GABA A receptor inhibitor, given five minutes before the end of strabismus surgery reduces the incidence of emergence agitation after sevoflurane anesthesia in children. Simultaneously, this study aims to find out the proper dose of midazolam with minimum disturbance to patient's emergence time.

DETAILED DESCRIPTION:
Sevoflurane is associated with a high incidence of emergence agitation in children. The etiology of emergence agitation is unclear. Some studies proposed that emergence agitation was related to a variable rate of neurologic recovery rate in different brain areas and immaturity of neurons. Inhalation anesthetics have been known to exert transient paradoxical excitatory effects in both animals and human patients, especially in children. The gamma(γ)-aminobutyric acid (GABA)A receptor is the target depressant effect site of most anesthetic drugs including sevoflurane. Midazolam acts on the benzodiazepine binding site of GABAA receptors and results in inhibitory effects on the central nervous system. The effect of midazolam premedication, as well as midazolam administration at the end of surgery, on suppressing emergence agitation has been studied. However, the effect of midazolam on emergence agitation is still controversial. This study aims to figure out the effect of midazolam at the end of surgery on emergence agitation during the recovery period, and find out the proper dose of midazolam with minimum disturbance to patient's emergence time.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists physical status I and II patients
* Aged one to 13 years scheduled to undergo strabismus surgery under general anesthesia
* Willing to be assigned to any of the study intervention groups

Exclusion Criteria:

* Refusal by parents
* Neurological disease
* Developmental delay
* History of any previous surgery
* Airway disease
* American Society of Anesthesiologists physical status score of III or IV

Ages: 1 Year to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Actual)
Dates: Start 2012-07; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Time of emergence | within the first 1hour after end of surgery
  The time of emergence is defined as time interval from the time of discontinuation of sevoflurane to the time of extubation.

SECONDARY OUTCOMES:
Incidence of emergency agitation | From just after extubation until the discharge of PACU, assessed up to 1 hour
  Agitation is assessed immediately after extubation, and continuously thereafter until participants are calm. Emergence agitation is evaluated using the four-point emergence scale and the pediatric anesthesia emergence delirium scale. The highest scores are recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Eun Jung Cho, Resident, Principal Investigator — Department of Anaesthesiology and Pain Medicine Department, Korea University Anam Hospital; S.Z. Yoon, Professor, Study Director — Department of Anaesthesiology and Pain Medicine Department, Korea University Anam Hospital
Locations (1):
- Department of Anaesthesiology and Pain Medicine Department; Korea University Anam Hospital, Seoul, South Korea